CLINICAL TRIAL: NCT06419192
Title: Evaluation of the Feasibility and Acceptability of Dietary Advice to Encourage Spontaneous Work: Randomised Pilot Study
Brief Title: Modifying Nutrition to Modify Delivery in Nulliparous Women
Acronym: MAMAN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DR230083
Record Dates: First submitted 2024-05-10; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Pregnant Woman
MeSH Terms: interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- dietary advice + food supplied (Experimental): Eat 7 dates a day from 37 weeks' gestation (SA) until delivery. Women will be provided with the quantity of dates they need.
  Interventions: Other: dietary advice; Other: food supplied
- dietary advice alone (Experimental): Advise to eat 7 dates a day from 37 weeks' gestation (SA) until delivery. The food will not be provided.
  Interventions: Other: dietary advice alone
- usual care (No Intervention): No specific dietary advice

INTERVENTIONS:
Other: dietary advice — Eat 7 dates a day from 37 weeks' gestation until delivery. Women will be provided with the quantity of dates they need.
  Arms: dietary advice + food supplied
Other: dietary advice alone — Advise to eat 7 dates a day from 37SA until delivery. The food will not be provided.
  Arms: dietary advice alone
Other: food supplied — Eat 7 dates a day from 37 weeks' gestation until delivery. Women will be provided with the quantity of dates they need.
  Arms: dietary advice + food supplied

SUMMARY:
In France, around 20% of women exceed the term of 41 weeks' amenorrhoea (SA). Maternal and foetal morbidity and mortality are increased when the term is exceeded, which justifies inducing labour. However, induction also increases maternal and foetal morbidity.

According to several studies, regular consumption of dates during the last month of pregnancy may increase the rate of spontaneous labour and natural childbirth.

Single-centre, randomised, open-label, 3-arm study :

Experimental group n°1: 'dietary advice + food provided'. Advice to eat 7 dates a day from 37 weeks' gestation until delivery. The quantity of dates required will be provided to the women.

Experimental group 2: 'dietary advice alone'. Advice to eat 7 dates a day from 37 weeks' gestation until delivery. The food will not be provided.

Control group: no specific dietary advice. Routine care group.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* Age ≥ 18 years
* Nulliparous
* Single pregnancy with fetus in cephalic presentation
* Pregnancy with physiological course
* Gestational age ≥ 34 and ⩽ 37 SA
* Membership of a social security scheme (CMU accepted)
* Signed informed consent

Exclusion Criteria:

* Any contraindication to vaginal delivery
* Presence of a foetal malformation
* Diabetes of any type (1, 2 or gestational)
* Food allergy contraindicating participation in the study
* Illiterate or non-French-speaking women
* Women under guardianship or trusteeship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 150 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Rate of compliance with dietary advice to eat 7 dates a day at the end of pregnancy in nulliparous women. | From 37 weeks'amenorrhoea to delivery (up to 41 weeks)

SECONDARY OUTCOMES:
Evaluation of women's experience of the intervention using a post-partum questionnaire | Following childbirth, during the stay in the maternity ward ; assessed up to 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Adeline DE WITT, MD, Study Director — University Hospital, Orléans
Locations (1):
- Gynaecology-obstetrics, University Hospital, Tours, Tours, France